CLINICAL TRIAL: NCT06325345
Title: A Randomized Controlled Trial of Gut-directed Hypnotherapy for Treatment of Irritable Bowel Syndrome in Ehlers-Danlos Syndromes and Generalized Hypermobility Spectrum Disorders
Brief Title: RCT of Gut-directed Hypnotherapy in Ehlers-Danlos Syndromes and Generalized Hypermobility Spectrum Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5277
Record Dates: First submitted 2023-02-08; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Ehlers-Danlos Syndrome; Irritable Bowel Syndrome; Hypermobility Syndrome; Gastrointestinal Dysfunction
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy (Other): Standard Medical Treatment will be administered by board certified gastroenterologists through the EDS Clinic gastroenterology clinical care pathway. Therapies will be individualized to the participants' current symptoms and severity of symptoms as per current clinical guidelines for management of IBS. Potential therapies that may be administered include dietary changes, supplemental fibre, and pharmacotherapy (including neuromodulators) as appropriate.
  Interventions: Other: Standard Medical Therapy
- Standard Medical Therapy plus Gut-Directed Hypnotherapy (Experimental): In addition to Standard Medical Therapy, participants randomized to this arm will attend 8 sessions of gut-directed hypnotherapy by a trained behavioral therapist. The treatment protocol developed for the proposed study was adapted from the empirically-supported Manchester Protocol for gut-directed hypnotherapy. At each visit, a voluntary, pleasant, and dream-like state of deep relaxation will be induced and suggestions made for greater relaxation, abdominal comfort, and normalization of gut function. The first session will be 90 minutes in duration and the remaining sessions will be 60 minutes. At the first session, participants will be provided with 30 minutes of education on the nature of the gut-brain axis and hypnotherapy before they undergo hypnotherapy.
  Interventions: Behavioral: Gut-directed hypnotherapy; Other: Standard Medical Therapy

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy — Eight session gut-directed hypnotherapy for IBS symptoms adapted from the evidence-based Manchester protocol for treatment of IBS.
  Arms: Standard Medical Therapy plus Gut-Directed Hypnotherapy
Other: Standard Medical Therapy — Standard medical treatment will be administered by board certified gastroenterologists

SUMMARY:
This randomized, controlled trial (RCT) will evaluate the effectiveness of gut-directed hypnotherapy for management of Irritable Bowel Syndrome (IBS) in individuals diagnosed with Ehlers-Danlos Syndromes or Generalized Hypermobility Spectrum Disorders (G-HSD). Consenting patients recruited from the Toronto General Hospital GoodHope Ehlers-Danlos Syndrome Clinic will be randomly assigned to one of two groups: (1) standard medical therapy or (2) standard medical therapy plus eight sessions of gut-directed hypnotherapy. The main questions this study will answer are:

1. Is gut-directed hypnotherapy an efficacious treatment for IBS symptoms among individuals with EDS or G-HSD?
2. Does gut-directed hypnotherapy improve other gut symptoms, quality of life, visceral sensitivity, and emotional distress?
3. Is the activity of the parasympathetic nervous system (i.e. the body's "rest and digest" system) associated with IBS symptoms or treatment outcomes among individuals with EDS or G-HSD?

All participants will be asked to meet with a gastroenterologist three times as part of the standard medical therapy. At each physician visit, they will undergo electrocardiogram recording and complete self-report measures of gastrointestinal symptoms, quality of life, visceral sensitivity, and emotional distress. Participants randomized to receive gut-directed hypnotherapy will also eight weekly remotely-delivered sessions of gut-directed hypnotherapy delivered by a trained behavioral therapist in between the first and second physician visit. At each session of gut-directed hypnotherapy, a voluntary, pleasant, and dream-like state of deep relaxation will be induced and suggestions made for greater relaxation, abdominal comfort, and normalization of gut function. The first session will also include 30 minutes of education on the nature of the gut-brain axis and hypnotherapy prior to hypnosis.

Researchers will compare study groups to see if participants who engaged in gut-directed hypnotherapy had greater improvement in IBS symptoms, other gastrointestinal symptoms, quality of life, visceral sensitivity, and emotional distress. Exploratory analyses will examine the relationships among heart rate variability, an index of parasympathetic nervous system activity, and study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Ehlers-Danlos Syndrome or Generalized Hypermobility Spectrum Disorder
* Physician diagnosis of Irritable Bowel Syndrome according to the Rome IV criteria.
* If receiving pharmacologic therapy for IBS, they must be on a stable dose for 4 weeks prior to study enrollment

Exclusion Criteria:

* Patients with diagnosed lower bowel disease (e.g. inflammatory bowel disease, celiac's disease)
* Patients with history of major gastrointestinal surgery (except appendectomy and/or cholecystectomy > 6 months prior to enrollment)
* Patients with limited comprehension of English or hearing difficulty who would not be able to understand the verbal instructions for clinical hypnosis
* Patients with a known history of serious mental illness (e.g., schizophrenia, dissociative identity disorder)
* Patients with cognitive deficits whose comprehension may limit benefit
* Patients with heavy alcohol use (> 15 drinks/week for men, > 10 drinks/week for women)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
IBS Symptom Severity | Immediately post-treatment, 3-months post-treatment
  The IBS Symptoms Severity Score (IBS-SSS) is a 5-item measure that asks participants to rate abdominal pain intensity, abdominal distension, dissatisfaction with bowel habits, and IBS life interference on a 0-100 scale. The IBS-SSS is a validated measure of IBS symptom severity and a recommended outcome measure for IBS treatment trials

SECONDARY OUTCOMES:
Upper Gastrointestinal Symptoms | Immediately post-treatment, 3-months post-treatment
  Upper gastrointestinal symptoms will be measured using the Patient Assessment of Upper Gastrointestinal Symptoms (PAGI-SYM), a commonly used 20-item self-report measure of upper gastrointestinal symptoms with good reliability and construct validity.
IBS-related Quality of Life | Immediately post-treatment, 3-months post-treatment
  IBS-related Quality of Life will be assessed using The Irritable Bowel Syndrome Quality of Life scale, a 34-item, psychometrically valid self-report measure of IBS-related QOL.
Visceral Sensitivity | Immediately post-treatment, 3-months post-treatment
  Visceral sensitivity will be evaluated by the Visceral Sensitivity Index (VSI). a 15-item measure developed to assess gastrointestinal specific anxiety. Visceral sensitivity has been identified as an important contributor to IBS symptom severity and a treatment target for IBS treatment. The VSI has excellent psychometric properties.
Emotional Distress | Immediately post-treatment, 3-months post-treatment
  Emotional Distress will be measured using the 8-item anxiety symptom and 8-item depressive symptom self-report measures from the Patient Reported Outcome Measurement Information System (PROMIS), which are extensively validated an have previously been used in IBS research.

OTHER OUTCOMES:
Weekly Ratings of GI Health and Medication Use | Once a week for 9 weeks hypnotherapy treatment
  Participants will rate upper abdominal pain, lower abdominal pain, abdominal distension, excess wind, disturbance in bowel movement, nausea, and vomiting on a scale from 0, no symptoms, to 10, severe symptoms. Participants will also rate their well-being over the past week on a scale from 0, no well-being, to 10, the most well-being possible. Participants will also be asked to report their opioid and cannabis use over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Liu, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No